CLINICAL TRIAL: NCT05841212
Title: The Acceptability and Feasibility of Implementing a Dialectical Behaviour Therapy (DBT) Skills Group for Adolescents with ADHD
Brief Title: DBT Skills Group for Adolescents with ADHD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRAS321708
Record Dates: First submitted 2023-03-16; First posted 2023-05-03 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DBT for ADHD (Other): The intervention will consist of a DBT skills group. Its name, length, style and content will be guided by the viewpoints shared in the intervention planning focus group/ individual interviews, and taken into consideration alongside a clinical rational and the evidence-based content. It will include skills from all four of the DBT modules: Mindfulness, Distress Tolerance, emotion regulation and interpersonal effectiveness. There will be an emphasis on the skills relevant to ADHD symptoms plus a core psychoeducational component on ADHD symptoms. The intervention will be adapted from Rathus and Miller's (2014) DBT for adolescents (DBT-A) manual.
  The group format will be didactic teaching with group discussion and experiential exercises to aid learning.
  Interventions: Other: DBT for ADHD

INTERVENTIONS:
Other: DBT for ADHD — See information included in arm/group description.

SUMMARY:
Attention Deficit Hyperactive Disorder (ADHD) is linked to three main symptoms: hyperactivity, inattention and impulsivity. It is increasingly being acknowledged that these symptoms have a wide-reaching impact on a person's life. Adolescents with ADHD are six times more likely to be excluded from school, have difficulties turn taking, express anger more often, have poorer emotion regulation and self-report a lower quality of life. In adulthood, people with ADHD are more likely to develop mental health difficulties, and to experience unemployment, divorce and be imprisoned. It is thought that emotion regulation and poor social skills are key factors leading to increases in mental health difficulties and poorer long term social outcomes. This pilot trial will look at whether an intervention which aims to increase emotion regulation and social functioning is acceptable and feasible. The intervention will be an adapted Dialectical Behaviour Therapy (DBT) skills group with an ADHD focus. DBT is an approach that aims to provide skills to assist an individual identify what they are feeling and change what they do in response to that feeling. For example, if an individual feels anger and the urge to be aggressive, DBT helps them to problem solve and find a more effective way of responding to their anger. Also, if an individual wants to communicate a relational need to others DBT helps them think about the most effective actions they can take to achieve this outcome. The intervention will be developed in collaboration with adolescents with ADHD. The intervention will then be delivered at the child and adolescent outpatient clinic site they received their diagnosis from. All participants will have a confirmed diagnosis of ADHD. Pre and post measures will be collected and reported on. The research team hope to commence recruitment in July 2023 and finish all data collection by 31st March 2024.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Attention Deficit Hyperactive disorder (using either DSM 5, DSM-IV, or ICD-10 - F90)
* Age 13-16 years
* Likely to benefit from DBT skills and can safely access/ engage in group interventions as assessed by clinical team [for intervention part]

Exclusion criteria:

* A low enough proficiency in written and spoken English that they would be unable to engage in the content of the group.
* Have not recently changed their medication in the last 2 weeks*, commenced a new medication in the last 2 weeks* or are receiving additional concurrent psychological intervention. (*calculated from the start of the intervention).
* The identified participant has recently taken part in another research trial and are at risk of research burden.
* Pose a risk to others in the group

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
25 participants with ADHD will be recruited from CAMHS services. | Within12-months
  To assess whether the intervention is feasible in terms of recruitment, for adolescents with ADHD.
60% of participants or more will attend all group sessions. | Within12-months
  To assess whether the intervention is feasible in terms of retention, for adolescents with ADHD.
60% or more of participants will complete a follow up measures. | Within12-months
  To assess whether the intervention is feasible in terms of retention, for adolescents with ADHD.
Individual participant attendance rate will be greater than 50%. | Within12-months
  To assess whether the intervention is feasible in terms of retention, for adolescents with ADHD.
66% of participants or more will report above neutral satisfaction ratings on weekly questionnaire | Within 12 months
  To assess whether participants will find both the intervention and assessment methods acceptable.
66% of participants or more from the focus group will report above neutral satisfaction. | Within 12 months
  To assess whether participants will find both the intervention and assessment methods acceptable, we will conduct a focus group and use thematic analysis to ascertain the satisfaction rating.

SECONDARY OUTCOMES:
At post-treatment compared to baseline participants will report improved levels of emotion regulation | Within 12 months
  Participants will complete the DERS-SF (2015) pre and post the intervention. We will report on any changes between baseline and post treatment score using effect sizes and confidence intervals. As this is a pilot trial tentative conclusions will be drawn from these findings.
At post-treatment compared to baseline participants will report a reduction in ADHD symptoms. | Within 12 months
  Participants will complete the Connors 3rd edition self report form and SNAP-IV-26 (1992) pre and post the intervention. We will report on any changes between baseline and post treatment score using effect sizes and confidence intervals. As this is a pilot trial tentative conclusions will be drawn from these findings.
At post treatment compared to baseline participants will report improved social skills and functioning. | Within 12 months
  Participants will complete the WSAS-Y (2019) pre and post the intervention. We will report on any changes between baseline and post treatment score using effect sizes and confidence intervals. As this is a pilot trial tentative conclusions will be drawn from these findings.
At post treatment compared to baseline participants will report improved social skills and functioning. | Within 12 months
  Participants will complete the SDQ (2005) pre and post the intervention. We will report on any changes between baseline and post treatment score using effect sizes and confidence intervals. As this is a pilot trial tentative conclusions will be drawn from these findings.

CONTACTS AND LOCATIONS:
Locations (1):
- South London and Maudsley Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.